CLINICAL TRIAL: NCT00901745
Title: Investigating the Interaction of Apelin and Angiotensin II Peripheral Resistance Vessels in Vivo in Man
Brief Title: Interaction of Apelin and Angiotensin in the Human Forearm Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Dr Gareth Barnes, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FS/09/019/26905 - 1b
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2009-05

CONDITIONS: Heart Disease; Vasodilation
Keywords: Renin angiotensin system; Apelin; Vasodilatation; Heart disease; Vascular biology
MeSH Terms: conditions — Heart Diseases; Aneurysm | interventions — Angiotensin II

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infusion of apelin (Experimental): Using forearm venous occlusion plethysmography apelin will be infused to cause reduction in forearm blood flow. Infusion of angiotensin II and noradrenaline will given and vasoconstriction will be assessed. Blood samples for the infused arm and contra-lateral arm will be taken at regular time points to assess local and systemic changes in relevant hormones.
  Interventions: Drug: Angiotensin II; Drug: Noradrenaline infusion
- Sodium nitroprusside infusion (Active Comparator): Using forearm venous occlusion plethysmography sodium nitroprusside will be infused to cause reduction in forearm blood flow. Infusion of angiotensin II and noradrenaline will given and vasoconstriction will be assessed. Blood samples for the infused arm and contra-lateral arm will be taken at regular time points to assess local and systemic changes in relevant hormones.
  Interventions: Drug: Angiotensin II; Drug: Noradrenaline infusion

INTERVENTIONS:
Drug: Angiotensin II — Infusion of up to 30picmol/ml angiotensin II will be infused and respondent vasoconstriction assessed.
Drug: Noradrenaline infusion — Infusion of up to 480 picomol/ml of noradrenaline will be infused.

SUMMARY:
The apelin-APJ system is a relatively new discovery. It has generated interest in part due to it's apparent ability to counteract the renin-angiotensin system, which is frequently overactive in many cardiovascular disease.

Apelin has the ability to cause blood vessels to relax, increasing their diameter and hence blood flow down the blood vessel. The researchers wish to investigate the hypothesis that an infusion of apelin will reduce the effects of angiotensin II, which is know to reduce the diameter of blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Healthy volunteers

Exclusion Criteria:

* Lack of informed consent
* Age < 18 years,
* Current involvement in other research studies,
* Systolic blood pressure >190 mmHg or <100 mmHg
* Malignant arrhythmias
* Renal or hepatic failure
* Haemodynamically significant aortic stenosis
* Severe or significant co morbidity
* Women of childbearing potential.
* Any regular medication

  * Previous history of any cardiovascular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in angiotensin II mediated vasoconstriction | 12 months

SECONDARY OUTCOMES:
Changes in relevant neurohumoral hormones in response to apelin infusion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gareth D Barnes, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Clincial Research Facility, Royal Infirmary of Edinburgh, 51 Little France Cresc, Edinburgh, United Kingdom